CLINICAL TRIAL: NCT04036006
Title: A National Trial of the ELM Lifestyle Program and Remission of the Metabolic Syndrome
Brief Title: Enhanced Lifestyles for Metabolic Syndrome
Acronym: ELM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Colorado, Denver (Other); Geisinger Clinic (Other); Rochester Institute of Technology (Other); University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Lynda Powell, PhD, MEd, Professor of Preventive Medicine, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18092408
Record Dates: First submitted 2019-04-18; First posted 2019-07-29 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Metabolic Syndrome
Keywords: Behavioral intervention; Lifestyle
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-Based (Experimental): The Group-based Program uses an ecologically valid setting in which participants exercise, prepare foods, and eat together to facilitate the emergence of old habits and replace them with healthy alternatives. The intervention team consists of a health psychologist, registered dietitian, and health coach. They co-facilitate group meetings for 15 participants that are held weekly for 3 months, bi-weekly for 3 months, and then monthly in participant-led maintenance meetings. Each session includes: weigh-in and physical activity (20 min), cooking demonstration (20 min), and a shared vegetable dish with discussion (50 min). The maintenance phase (months 7 to 24 post randomization) consists of support and health-related topics of the participants' own choosing. Progress reports with lab results are sent to participants and primary care physicians.
  Interventions: Behavioral: Group-Based Program
- Self-Directed (Active Comparator): The Self-Directed lifestyle program represents enhanced usual care based upon what is currently offered in primary care in the United States for lifestyle treatments for adults with metabolic syndrome. Usual care is enhanced by: 1) lifestyle education for management of metabolic syndrome provided in evidence-based tip sheets from nationally recognized organizations; 2) provision of a Fitbit for self-monitoring physical activity; 3) access to a website containing all education materials; and 4) progress report letters with lab results sent to participants and primary care physicians after completion of each assessment
  Interventions: Behavioral: Self-Directed Program

INTERVENTIONS:
Behavioral: Group-Based Program — The Group-based Program uses an ecologically valid setting in which participants exercise, prepare foods, and eat together to facilitate the emergence of old habits and replace them with healthy alternatives. The intervention team consists of a health psychologist, registered dietitian, and health coach. They co-facilitate group meetings for 15 participants that are held weekly for 3 months, bi-weekly for 3 months, and then monthly in participant-led maintenance meetings. Each session includes: weigh-in and physical activity (20 min), cooking demonstration (20 min), and a shared vegetable dish with discussion (50 min). The maintenance phase (months 7 to 24 post randomization) consists of support and health-related topics of the participants' own choosing. Progress reports with lab results are sent to participants and primary care physicians.
  Arms: Group-Based
Behavioral: Self-Directed Program — The Self-Directed lifestyle program represents enhanced usual care based upon what is currently offered in primary care in the United States for lifestyle treatments for adults with metabolic syndrome. Usual care is enhanced by: 1) lifestyle education for management of metabolic syndrome provided in evidence-based tip sheets from nationally recognized organizations; 2) provision of a Fitbit for self-monitoring physical activity; 3) access to a website containing all education materials; and 4) progress report letters with lab results sent to participants and primary care physicians after completion of each assessment.
  Arms: Self-Directed

SUMMARY:
This is a multi-center behavioral randomized trial with the aim of comparing a group-based lifestyle intervention with a self-directed lifestyle intervention on remission of the metabolic syndrome over 2 years of follow-up.

DETAILED DESCRIPTION:
The purpose of this trial is to determine the efficacy and cost-effectiveness of the Group-Based and Self-Directed ELM lifestyle programs when offered on a national level. A multi-site randomized trial will be conducted on 600 patients with the metabolic syndrome (MetS) by five national sites, each of which will randomize 120 patients to the Group-Based or Self-Directed programs. The Group-Based program targets healthy eating, physical activity, and stress reduction and is based upon neuroscience studies showing that mindful habits provide resilience against the power of emotions to subvert intention, and social science studies showing that sustainability is enhanced by support from a health network. The Self-Directed program represents enhanced usual care based upon what is currently offered in medicine and wearable technology for treatment of adults with MetS and its components. The primary outcome is remission of MetS at 2 years. Secondary outcomes include cost-effectiveness, vegetable intake, physical activity, and mindful awareness.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with metabolic syndrome, defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO (Alberti, 2009). Note that hemoglobin A1c will be measured as a marker of impaired glucose metabolism, but will not be considered in determining metabolic syndrome status. To meet metabolic syndrome criteria the participant should have ≥ 3 of the following five criteria:

   * Waist circumference based on AHA/NHLBI (ATP III) cut points of ≥ 102 cm for men and ≥ 88 cm for women
   * Fasting triglycerides ≥150 mg/dL or treatment for elevated triglycerides
   * Fasting HDL cholesterol <40 mg/dL in men or <50 mg/dL in women, or treatment for low HDL
   * Systolic blood pressure ≥130 m Hg, diastolic blood pressure ≥85 mm Hg, or treatment for hypertension
   * Fasting plasma glucose 100-125 mg/dL (range inclusive)
2. Greater than 18 years of age

Exclusion Criteria:

1. Unable to walk 2 consecutive blocks without assistance, based on patient report.
2. Unwilling, unable, or not ready to make the lifestyle changes prescribed in ELM
3. Unwilling to be randomized to either arm of the trial
4. Unable or unwilling to give an informed consent, communicate with study staff, or complete the study run-in period. The run-in period requires attending an information session, completing two assessment visits within the scheduled time (potential participant is allowed to reschedule once), wearing an accelerometer, and completing lifestyle logs (see protocol)
5. Does not have reliable access to the internet via a computer or mobile device
6. Not fluent in English
7. Current diagnosis of type 1 or type 2 diabetes, or on any diabetes medications except metformin
8. Inpatient treatment for a psychiatric condition within the past 6 months, or currently receiving treatment for schizophrenia or other serious psychiatric illness
9. Probable major depression, defined as a PHQ-8 score ≥10
10. Pregnant women, planning a pregnancy in the next 24 months, given birth in the last 6 months, or currently breastfeeding
11. ≥ 30 total days of oral corticosteroid use within the last year, history of solid organ transplant, or history of stem cell transplant
12. Problematic use of alcohol and/or recreational drugs based on the ASSIST screening tool (score of ≥27).
13. Self-reported or known history of an eating disorder (e.g., binging and purging) in the past 5 years
14. Use of weight loss medications (Qsymia, phentermine, etc.) or supplements in the last 3 months, or unwilling to abstain from taking weight loss medications or supplements during the study
15. History of bowel resection surgery or bariatric surgery
16. Participant does not have, or is unwilling to seek care from, a primary care physician at the time of enrollment
17. Any medical condition known to influence the etiology of MetS as judged by the study physician (e.g., uncontrolled hypothyroidism, endocrine hypertension, etc)
18. History of major cardiovascular illness, including a) stroke; b) myocardial infarction; c) congestive heart failure requiring hospitalization, or greater than NYHA heart failure class I; d) uncontrolled hypertension (SBP>180 or DBP > 105); e) unstable angina; or f) other major cardiovascular illness which the site PI determines could limit ability to participate in the trial.
19. Behavioral/logistical barriers to trial participation or engagement, e.g., a scheduled major surgery, scheduling difficulties, travel plans, moving outside the study area
20. Cognitive impairment, defined by a Montreal Cognitive Assessment (MoCA) score of ≤25. The MoCA will be administered only when research staff suspect cognitive impairment
21. Visual or hearing impairment
22. Severe food allergies or food intolerances/preferences that preclude participation in the ELM program
23. Currently taking or expecting to take any of the following exclusionary medications:

    1. Antiretroviral therapy (e.g., HAART)
    2. Weight loss medications (as in #14)
    3. Medications known to significantly influence weight or metabolic outcomes
    4. Diabetes drugs other than metformin (as in #7)
24. Participation in any clinical trial, until at least six months following the end of the intervention phase. Individuals in long-term follow-up (over 6 months post intervention) may be enrolled in ELM.
25. Cancer treatment within the last 6 months, excluding chemoprophylaxis or treatment for non-melanoma skin cancer.
26. Previous participation in an ELM program or currently living with ELM participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Remission of Metabolic Syndrome | Measured at 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the proportion of participants who are in remission of the metabolic syndrome (MetS) at 2 years. MetS is defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO as having 3 or more risk factors for cardiovascular disease. To be considered in remission of MetS the participant must have less than 3 of the following 5 criteria: 1) Waist circumference based on AHA/NHLBI (ATP III) cut points of ≥ 102 cm for men and ≥ 88 cm for women; 2) Fasting triglycerides ≥150 mg/dL or treatment for elevated triglycerides; 3) Fasting HDL cholesterol <40 mg/dL in men or <50 mg/dL in women, or treatment for low HDL; 4) Systolic blood pressure ≥130 m Hg, diastolic blood pressure ≥85 mm Hg, or treatment for hypertension; and 5) Fasting plasma glucose 100-125 mg/dL.
  Analysis will be performed on pre-determined subgroups: education, sex, site, weight, BMI, MetS severity, race, income # of comorbidities, self-efficacy, and age.

SECONDARY OUTCOMES:
Vegetable consumption | Measured at 6, 15, and 24 months following treatment assignment
  Compare the Group-Based and Self-Directed arms on the proportion of participants who eat 2 cups of vegetables per day. This will be assessed using the National Cancer Institute (NCI) Fruit and Vegetable Intake Screener from the Eating at America's Table Study: All Day Screener.
Physical activity | Measured at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the proportion of participants who achieve 150 minutes of at least moderate intensity physical activity per week. Activity is measured using an accelerometer (Actigraph wGT3X-BT) worn on the right hip for 7 days and for at least 10 hours/day.
Facets of Mindfulness | Measuring change from baseline mindfulness at 6, 15, and 24 months following treatment assignment.
  Participants will complete the Five Facet Mindfulness Questionnaire. A subscale comprised of 3-facets (observe, act with awareness, and nonreact) will be utilized to measure mindfulness in ELM. Group-Based and Self-Directed arms will be compared on the proportion of participants who improve in a 3-facet mindfulness score of greater than or equal to 1 standard deviation of baseline distribution. The scale range for the 5-facet mindfulness questionnaire is 39-195 with a lower score reflecting less mindfulness. The 3-facet scale range is 23-115 with a lower score reflecting less mindfulness.
Habit formation | Measuring at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the proportion of participants who improve in habit strength in 4 domains (diet, physical activity, emotional control, and sensory awareness), defined as a mean of ≥ 4 on the Self-Report Habit Index. A 5-point Likert scale will be used with a scale range from 0 to 20. A lower score reflects a weaker habit.
Cost-effectiveness | Measured over the 24 month patient participant follow-up period
  Calculate the cost-effectiveness of the Group-Based relative to the Self-Directed programs. Cost-effectiveness will be be quantified by using the Incremental Cost-Effectiveness Ratio and will reflect the additional cost of the Group-Based program relative to the Self-Directed Program in its efficacy at promoting a sustained remission of metabolic syndrome.
Healthcare utilization | Measured over the 24 month patient participant follow-up period
  Compare the Group-Based and Self-Directed programs on health care utilization (primary care visits, specialty care visits, ER visits, hospital admissions). Participants are queried quarterly concerning use of health care services.
Cost of Medications | Measured at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed programs on the cost of prescribed medications. This will include collecting data on the number of prescribed medications including data on the number of medications and dosage (mg) of each medication.
Number of Prescribed Medications | Measured at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed programs on the number of prescribed medications self-reported by participants.
Severity of Metabolic Syndrome | Measured at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the severity of the Metabolic Syndrome (MetS). MetS components will be assessed as a continuous sex- and race/ethnicity-specific score (Gurka MJ, Lilly CL, Oliver MN, DeBoer MD. An examination of sex and racial/ethnic differences in the metabolic syndrome among adults: a confirmatory factor analysis and a resulting continuous severity score. Metabolism. 2014;63:218-25).
Weight Loss | Measuring change from baseline at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on average weight loss (kg). Weight is recorded in kilograms to the nearest 0.1 kg using a flat scale.
≥ 5% body weight loss | Measuring change from baseline at 6,15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the proportion of participants with ≥ 5% loss of baseline weight (kg). Weight is recorded in kilograms to the nearest 0.1 kg using a flat scale.
Body Mass Index | Measured at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on Body Mass Index (BMI). Height will be recorded in cm to nearest 0.25 cm and weight recorded in kg to nearest 0.1 kg. BMI = weight (kg) / height squared (m)
Blood Pressure (metabolic syndrome component) | Measured at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the blood pressure component of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. The criteria for blood pressure is met when systolic blood pressure ≥130 m Hg, diastolic blood pressure ≥85 mm Hg, or self-reported treatment for hypertension.
  Average of 3 seated resting blood pressure measurements using NHANES protocol and cuff sizes based on arm circumference. Device is OMRON HEM-907XL
  Cuff sizes:
  Small (17.0-22.0 cm) Medium/Adult (22.1-32.0 cm) Large (32.1-42.0 cm) Extra Large (42.0-50.0 cm)
Waist Circumference (metabolic syndrome component) | Measured at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the waist circumference component of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. The criteria is based on AHA/NHLBI (ATP III) cut points of ≥ 102 cm for men and ≥ 88 cm for women.
  Waist circumference will be measured using a tape measure, following the National Heart, Lung, and Blood Institute waist circumference assessment guidelines.
Triglycerides (metabolic syndrome component) | Measured at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the triglyceride component of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. The criteria for elevated triglyceride levels are fasting triglycerides ≥150 mg/dL or treatment for elevated triglycerides.
  A fasting blood sample will be sent to Quest diagnostics for analysis.
High-Density Lipoproteins (HDL) Cholesterol (metabolic syndrome component) | Measured at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the HDL cholesterol component of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. The criteria for low HDL are fasting HDL cholesterol <40 mg/dL in men or <50 mg/dL in women, or treatment for low HDL.
  A fasting blood sample will be sent to Quest diagnostics for analysis.
Fasting Plasma Glucose (metabolic syndrome component) | Measured at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on each of the five components of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. Fasting plasma glucose 100-125 mg/dL (range inclusive) is considered a component of the metabolic syndrome. A fasting blood sample will be sent to Quest diagnostics for analysis.
Frequency of Contacts within Health network | Measuring change from baseline at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the frequency of contacts within participants' health network.
Energy and vitality Index | Measured at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on the energy and vitality subscale from the Medical Outcomes Study 36-item Short-Form Health Survey (SF-36) version 1. The scale range is 0 to 100 with a low score reflecting a lower energy and vitality.
Perceived stress | Measuring change from baseline at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on change of perceived stress score from baseline using the 10-item Perceived Stress Scale. The scale range is from 0 to 40. A lower score reflects lower levels of stress.
Depressive symptoms | Measuring change from baseline at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on change of depressive symptoms from baseline using the 8-item self-report Patient Health Questionnaire Depression Scale (PHQ-8). This scale ranges from 0 to 24 with a lower score reflecting less (or no) depressive symptoms.
Social support for diet | Measured at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on social support for diet. The Social Support for Diet Survey assesses the level of support individuals making health-behavior changes (eating habits) feel they receive from family and friends. This scale is divided into two subscales: 1) encouragement from family and friends and 2) discouragement from family and friends. The Encouragement subscale ranges from 5 to 25 with a lower score reflecting less encouragement (negative outcome). The Discouragement subscale ranges from 5 to 25 with a lower score reflecting less discouragement (positive outcome).
Social support for exercise | Measured at 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on social support for exercise. The Social Support for Exercise Survey assesses the level of support individuals making health-behavior changes (exercise) feel they receive from family and friends. This questionnaire includes two subscales: 1) Participation and 2) Family Rewards and Punishment. The Participation subscale ranges from 10-50 with a low score reflecting less participation of family and friends (negative outcome). The Family Rewards and Punishment subscale ranges from 3 to 15 with a lower score reflecting increased family rewards (positive outcome).
Hemoglobin A1c levels | Measured at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on Hemoglobin A1c levels. A blood assay will be analyzed by Quest Diagnostics. Standard safety procedures are used in performing the participant blood draw required for this measure.
Sugar-sweetened beverages | Assessed during in-person participant assessments conducted at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on frequency of consumption of sugar-sweetened beverages using the Behavioral Risk Factor Surveillance System - Beverage Items.
Eating competence | Measured at baseline and 6, 15, and 24 months following treatment assignment.
  Compare the Group-Based and Self-Directed arms on eating competence using the 16-item Eating Competence Survey. The scale ranges from 0 to 48 with a higher score reflecting a better outcome.
Impact of pandemic | Measured at 24 months following treatment assignment.
  Compare results between participants in Wave 1 and those in Waves 2, 3, & 4. on the primary outcome at 2 years. MetS is defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO as having 3 or more risk factors for cardiovascular disease. To be considered in remission of MetS the participant must have less than 3 of the following 5 criteria: 1) Waist circumference based on AHA/NHLBI (ATP III) cut points of ≥ 102 cm for men and ≥ 88 cm for women; 2) Fasting triglycerides ≥150 mg/dL or treatment for elevated triglycerides; 3) Fasting HDL cholesterol <40 mg/dL in men or <50 mg/dL in women, or treatment for low HDL; 4) Systolic blood pressure ≥130 m Hg, diastolic blood pressure ≥85 mm Hg, or treatment for hypertension; and 5) Fasting plasma glucose 100-125 mg/dL.
  Analysis will be performed on pre-determined subgroups: education, sex, site, weight, BMI, MetS severity, race, income # of comorbidities, self-efficacy, and age.

OTHER OUTCOMES:
Pre-specified outcomes | Measured at 24 months after treatment assignment.
  To evaluate the impact of ELM lifestyle programs on reversing the metabolic syndrome for specific subgroups. These subgroups include: education, sex, site, weight, BMI, metabolic syndrome severity, race, income, number of comorbidities, self-efficacy, and age.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Powell, PhD, Study Chair — Rush University Medical Center; Sumihiro Suzuki, PhD, Study Director — Rush University Medical Center
Locations (5):
- United States (5):
  - CU Anschutz Health and Wellness Center, Aurora, Colorado
  - Department of Family and Preventive Medicine, Rush University Medical Center, Chicago, Illinois
  - University of Missouri-Kansas City, Kansas City, Missouri
  - Rochester Institute of Technology, Rochester, New York
  - Geisinger, Danville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Powell LH, Berkley-Patton J, Drees BM, Karavolos K, Lohse B, Masters KS, Nicklas JM, Rothschild SK, Yeh C, Zimmermann LJ, Suzuki S; ELM Trial Research Group. Lifestyle Intervention for Sustained Remission of Metabolic Syndrome: A Randomized Clinical Trial. JAMA Intern Med. 2026 Jan 1;186(1):67-77. doi: 10.1001/jamainternmed.2025.5900. PMID 41207299
- [Derived] Yeh C, Crane MM, Daniels B, Lohse B, Karavolos K, Olinger T, Nicklas J, Powell LH, Suzuki S. Factors associated with male recruitment in a multi-site randomized behavioral clinical trial targeting the metabolic syndrome: analysis of screening and recruitment data from the ELM trial. Trials. 2024 Dec 21;25(1):844. doi: 10.1186/s13063-024-08703-8. PMID 39707544

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT04036006/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT04036006/ICF_002.pdf